CLINICAL TRIAL: NCT03488381
Title: Effects of Repetitive Subconcussive Head Impacts on Ocular-motor Function and Brain-derived Blood Biomarker
Brief Title: Effects of Soccer Heading on Ocular-motor Function and Blood Biomarker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Keisuke Kawata, Assistant Professor of Kinesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1610743422
Record Dates: First submitted 2018-03-20; First posted 2018-04-05 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Trauma, Head
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soccer Heading (Experimental)
  Interventions: Device: Soccer Heading
- Kicking-Control (Sham Comparator)
  Interventions: Device: Soccer Heading

INTERVENTIONS:
Device: Soccer Heading — Soccer Heading: Subjects stood approximately 40 feet away from a JUGS soccer ball launcher and participated in 10 consecutive soccer headings, separated by one minute intervals.
  Soccer Kicking: Subjects stood approximately 40 feet away from a JUGS soccer ball launcher and participated in 10 consecutive soccer kicks, separated by one minute intervals.
  Other Names: Soccer Kicking

SUMMARY:
Repetitive head impacts in sports and military may cause deleterious effects in the nervous system. Investigators' previous works in football players have shown promising results in prediction of concussion and prevention of long-term defect using eye-movement paradigm (ocular-motor system) and blood biomarker. However, acute head impact effects on aforementioned parameters remain unknown. Thus, to answer a critical research question that whether or not ocular-motor system and brain-derived blood biomarker may be acutely altered following 10 successions of controlled soccer heading. To answer the question, investigators hypothesized that acute bout of soccer heading will not elicit noticeable change in subject's symptoms but to induce a transient defect in the ocular-motor system and increase plasma expression of brain-derived biomarker.

DETAILED DESCRIPTION:
Adult aged soccer players aged 18-26 years will be recruited via listserv email to Indiana University undergraduate students. Once subjects fulfill inclusion criteria and free of exclusion criteria, participants will be randomly assigned to one of two groups (Heading vs. Kicking).

For non-athletic control cohort, investigators will attempt to recruit 20 subjects who are 18-26 years old, have never played organized sports, and have never been diagnosed with a concussion before. This cohort is to evaluate and account for the soccer players' baseline, which may be influenced by a history of repetitive heading and sports participation. This group will participate in a single test session that lasts approximately in 1.5 hours. During the session, blood draw (4mL, about 1 teaspoon), measure eye movements using an ocular motor headset,

The study consists of 4 data collection time points in a 2-day period. This study design will enable to test outcome measures over 3 acute phases.

* The 1st test session takes place right before the intervention (soccer heading or kicking).
* Participants will perform either soccer heading or kicking.
* The 2nd test session takes place right after the intervention (soccer heading or kicking).
* The 3rd test session takes place 2h after the intervention (soccer heading or kicking).
* The 4th test session takes place approximately 24h after the intervention.

A standardized and reliable soccer heading protocol will be used for the experiment. A triaxial accelerometer (Triax Technologies) embedded in a head-band pocket and positioned back of the head to monitor linear and rotational head accelerations. A JUGS soccer machine will be used to simulate a soccer throw-in with a standardized ball speed of 25mph across both groups. Soccer players frequently perform this maneuver during practice and game. Subjects will stand approximately 40ft away from the machine to perform either the heading or kicking. Participants in the heading group perform 10 standing headers with 1 header per minute, whereas kicking control group performs 10 kicks. The participants in the heading and kicking groups will be instructed to direct the ball back toward the JUGS soccer machine in the air.

During each test session, various assessments will be conducted on each subject. First, the post-concussion symptom scale, as a subset of the Sports Concussion Assessment Tool 3, will be used as a method of assessing the presence and severity of symptoms. This paper-pencil symptom checklist consists of 22 symptoms with 7-point Likert scale per symptom to monitor subject's well-being. Next, Antecubital vein blood draws will be performed each test session to help determine blood biomarker concentrations. A certified phlebotomist will thoroughly clean the elbow surface with an alcohol swab and draw 4 ml of whole blood (approx. 1 teaspoon) into vacutainer tubes containing EDTA anti-coagulant with 21G butterfly needle. A Total of 16 ml blood for the study (4 ml x 4 time points; 3~4 teaspoons). After the blood draw, the subject will use gauze to maintain direct pressure for 3 mins and Band-Aid will be provided. The whole blood will be centrifuged at 3,000 revolutions per minute for 20 minutes at 4°C after 40 mins of coagulation. The plasma will then be divided and transferred into 1 mL cryovials and flash frozen and stored at -80°C in Exercise Biochemistry lab.

The subject will then perform eye-movement tasks using the EYE-SYNC headset. This visual-tracking protocol has been replicated and validated in a number of concussion and sleep deprivation studies, however to investigators' knowledge this study for the first time will unravel subconcussive effects. Prior to testing, a Snellen chart will be used to verify that the subject has a normal or corrected-to-normal vision (minimum 20/30). The subject will be seated in a normally lit room and stabilize the headset with two hands while the elbows placed on the desk. The visual stimulus will be presented using a 120-Hz frame rate LCD screen in the headset and binocular eye movements will be tracked by a single camera secured in the headset. The test stimulus consists of a red circular target, 0.5° diameter in a visual angle with a 0.2° black dot in the center. The target moves in a circular clockwise trajectory of 10° radius at 0.4 Hz, with the target speed corresponding to 25°/s. The entire testing sequence will last approximately 3 mins consisted of a calibration and 2 consecutive test runs. Calibration of the eye position is conducted by having the subject fixate on a target presented at eight locations on the circular path of the test stimulus and one additional fixation point at the center of the circular path. The fixation target was presented at these nine locations in a randomized order. Each of the two test runs consists of 6 cycles of circular movement corresponding to 15 s in duration per test run. The subject will be instructed as "follow the movement of the target as closely as possible."

ELIGIBILITY:
Inclusion Criteria:

For Soccer Cohort

1. being between 18 to 26 years of age
2. an active member of a soccer team (i.e., collegiate, intramural, club, professional)
3. at least 5 years of soccer heading experience.

For non-Athletic Control Cohort

1. Being between 18 to 26 years of age
2. Have never played organized sports
3. Have never been diagnosed with a concussion

Exclusion Criteria:

For both Soccer and Non-Athletic Control cohorts

1. any head, neck, or face injury in the 1 year prior to the study (e.g., concussion, eye injury);
2. history of vestibular, ocular, or vision dysfunction (e.g., macular degeneration)
3. currently taking any medications affecting balance (e.g., antibiotics)
4. pregnancy
5. HIV
6. any neurological disorders (e.g., seizure disorders, closed head injuries with loss of consciousness greater than 15 minutes, CNS neoplasm, spinal cord injury/surgery, history of stroke)
7. hypertension, cardiac arrhythmia, or pulmonary disease
8. lower extremity injury that would prohibit normal walking
9. metal implants in the head
10. implantation of cochlear device, cardiac pacemaker, medical fusion device, intracardiac lines, or neurostimulator (e.g., DBS, epidural/subdural VNS)
11. history of severe injury to the bones, joints, or muscles in either arm

    Session-specific exclusion criteria will include:
12. slept less than 4 hours before the 1st and 2nd test day (verified by the TMS screening questionnaire)
13. drank more than 3 alcoholic drinks or used recreational drugs 24 hours before the 1st and 2nd test day
14. drank more than 3 cups of coffee in an hour before test sessions
15. glasses are prohibited (contact lens are okay) for safety purpose for the heading intervention

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Changes in Brain-Derived Blood Biomarker Over Time in Relation to the Baseline | Measured at four time points (pre-intervention, immediately post-intervention, 2 hours post, and 24 post)
  Outcome measure will be the slope of increased (worsened) levels of blood biomarkers compared to the baseline and control group
Changes in Ocular-Motor Function Over Time in Relation to the Baseline | Measured at four time points (pre-intervention, immediately post-intervention, 2 hours post, and 24 post)
  Outcome measure will be the slope of increased (worsened) levels of ocular-motor performance compared to the baseline and control group

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States

REFERENCES:
- [Derived] Huibregtse ME, Nowak MK, Kim JE, Kalbfell RM, Koppineni A, Ejima K, Kawata K. Does acute soccer heading cause an increase in plasma S100B? A randomized controlled trial. PLoS One. 2020 Oct 23;15(10):e0239507. doi: 10.1371/journal.pone.0239507. eCollection 2020. PMID 33096545
- [Derived] Huibregtse ME, Ejima K, Chen Z, Kalbfell RM, Koppineni A, Kawata K. Acute Time-Course Changes in CCL11, CCL2, and IL-10 Levels After Controlled Subconcussive Head Impacts: A Pilot Randomized Clinical Trial. J Head Trauma Rehabil. 2020 Sep/Oct;35(5):308-316. doi: 10.1097/HTR.0000000000000597. PMID 32881764
- [Derived] Nowak MK, Bevilacqua ZW, Ejima K, Huibregtse ME, Chen Z, Mickleborough TD, Newman SD, Kawata K. Neuro-Ophthalmologic Response to Repetitive Subconcussive Head Impacts: A Randomized Clinical Trial. JAMA Ophthalmol. 2020 Apr 1;138(4):350-357. doi: 10.1001/jamaophthalmol.2019.6128. PMID 32053162

DOCUMENTS (2):
  • Study Protocol (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT03488381/Prot_000.pdf
  • Informed Consent Form (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT03488381/ICF_001.pdf